CLINICAL TRIAL: NCT06615193
Title: A Phase Ia/Ib, Open-label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HDM2005 in Patients With Relapsed/Refractory B-cell Lymphoma and Advanced Solid Tumor
Brief Title: A Study of HDM2005 in Patients With Relapsed/Refractory B-cell Lymphoma and Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HDM2005-101
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumors; Refractory Lymphoma; Relapsed Hematologic Malignancy
MeSH Terms: conditions — Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HDM2005 (Experimental): In dose escalation phase, participants will be administered escalating doses of HDM2005 at 0.3~2.75mg/kg IV on Day 1 of repeated 21-day cycles.
  In dose expansion phase, participants will be administered to recommended dose for expansion (RDE) of HDM2005 on Day 1 of repeated 21-day cycles .
  Interventions: Drug: HDM2005

INTERVENTIONS:
Drug: HDM2005 — HDM2005 will be administered via IV infusion.

SUMMARY:
This is a first-in-human (FIH) study to evaluate the safety and preliminary efficacy of experimental drug HDM2005 in patients with relapsed/refractory B-cell lymphoma and advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the study treatment protocol and visit schedule, enroll voluntarily and sign a written informed consent;
2. Male or female aged ≥ 18 years at the time of signing the ICF;
3. B-cell lymphoma: ECOG performance status of 0-2;
4. Advanced solid tumors: ECOG performance status of 0-1;
5. Life expectancy of at least 3 months;
6. Dose escalation phase: Histopathologically confirmed relapsed/refractory B-cell lymphoma following at least 2 prior lines of systemic therapy;
7. Dose expansion phase: relapsed/refractory B-cell lymphoma and advanced or metastatic solid tumor of specified type.
8. All subjects are required to provide archived tissue (5 unstained sections) obtained within the previous 2 years or fresh tissue for ROR1 expression testing at the central laboratory; in addition, relapsed/refractory lymphoma subjects are required to provide tissue sections used for previous pathological diagnosis for pathological consultation at the central laboratory;
9. Relapsed/refractory B-cell lymphoma: Subjects in Phase Ia dose escalation phase should have evaluable lesions; subjects in Phase Ib dose expansion phase should have at least 1 radiographically measurable lymph node or extranodal malignant tumor lesion (intranodal lesion defined as having a long diameter > 1.5 cm; extranodal lesion having a long diameter > 1.0 cm) as assessed by computed tomography (CT)/magnetic resonance imaging (MRI) according to 2014 Lugano criteria, and a lesion that has previously received radiotherapy is considered measurable when it shows unequivocal progression after completion of radiotherapy;
10. Advanced solid tumors: subjects are required to have at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 ;
11. Subjects must have recovered (to ≤ Grade 1) from any AE associated with prior anticancer therapy;
12. Subjects have adequate organ and bone marrow function;
13. Female subjects of childbearing potential should agree to use contraception methods (e.g., intrauterine device, contraceptive pill, or condom) during the study and for 6 months after the end of the study; have a negative serum pregnancy test within 7 days before study enrollment; and male subjects should agree to use contraceptive avoidance measures during the study and for 6 months after the end of the study.

Exclusion Criteria:

1. B-cell lymphoma: known central nervous system (CNS) involvement .
2. Advanced solid tumors: Patients with active brain metastases (defined as stable for < 4 weeks, or symptomatic, or requiring antiepileptic drug/hormonal therapy, or meningeal metastases);
3. Subjects with prior allogeneic HSCT who have developed acute graft-versus-host disease (GVHD) or persistent evidence of chronic GVHD (as manifested by ≥ Grade 2 serum bilirubin, ≥ Grade 3 skin involvement, or ≥ Grade 3 diarrhea or receiving systemic immunosuppressive therapy/prophylaxis for GVHD);
4. Subjects have another primary malignancy ,with the following exceptions: adequately treated non-melanoma skin cancer without evidence of disease recurrence and adequately treated carcinoma in situ without evidence of disease recurrence,et al;
5. History of severe bleeding disorders ;
6. History of chronic pancreatitis or acute pancreatitis within 6 months;
7. History of interstitial lung disease, radiation pneumonitis requiring steroid therapy, or any evidence of clinically active interstitial lung disease;
8. Patients with uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage after intubation and drainage, VEGF inhibitors, platinum and other drugs injection (subjects with stable symptoms for at least one week after treatment can be enrolled);
9. Prior solid organ transplantation;
10. Persistent peripheral neuropathy > Grade 1 at baseline;
11. Clinically significant cardiovascular or cerebrovascular diseases;
12. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection requiring systemic therapy (except for localized skin or nail bed fungal infection) at enrollment;
13. Active infectious disease, such as HIV infection, active hepatitis B, active hepatitis C (positive RNA result), active syphilis;
14. Receiving corticosteroids (prednisone equivalent more than 30 mg/day);
15. Contraindication to any component of HDM2005;
16. History of drug anaphylactic shock, severe food allergy, uncontrolled asthma/COPD;
17. Female subjects who are pregnant, lactating or planning to become pregnant during the study;
18. Known history of mental illness or substance abuse that would impair the subject's ability to cooperate with study requirements;
19. Prior or current evidence of any disease, treatment, or laboratory abnormality that, in the opinion of the investigator, could affect the outcome of the study, prevent the subject from participating in the study entirely, or is not in the subjects' best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events (for dose escalation phase) | up to 21 days following first dose
  DLT will be determined by definition during the DLT observation period.
Incident and severity of adverse events(for dose escalation phase) | Until 28 days after the last dose or initiation of a new antineoplastic therapy, whichever occurs first
  The safety profile of HDM2005 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Objective Response Rate (ORR)(for dose expansion phase) | Until withdrawal of consent, loss to follow-up, initiation of other new antineoplastic therapy, end of study, or study termination by the sponsor, whichever occurs first (up to approximately 3.5 years)
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the investigator.
Recommended Phase 2 Dose (RP2D) (for dose expansion phase) | Approximately 3.5 years
  The selection of RP2D will be based on consideration of overall safety information together with available pharmacokinetic,E-R relationships, and efficacy data.

SECONDARY OUTCOMES:
Plasma concentration of HDM2005, total antibody and the free MMAE | up to 28 days following last dose
  Plasma concentration of HDM2005, total antibody and the free MMAE will be reported for each arm.
Immunogenicity | up to 28 days following last dose
  Number and percentage of anti-drug antibody (ADA)-positive patients will be assessed.
Incident and severity of adverse events(for dose expansion phase) | Until 28 days after the last dose or initiation of a new antineoplastic therapy, whichever occurs first
  The safety profile of HDM2005 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Objective Response Rate (ORR)(for dose escalation phase) | Approximately 3.5 years
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the investigator.
Time to Response (TTR) | Approximately 3.5 years
  TTR is defined as the interval from the start of study therapy to the first documentation of an objective response.
Progression free survival (PFS) | Approximately 3.5 years
  PFS is defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression/relapse or death from any cause.
Duration of Response (DOR) | Approximately 3.5 years
  DOR is defined as the interval from the first documentation of objective response to the earlier of the first documentation of disease progression/relapse or death from any cause.
Overall survival (OS) | Approximately 3.5 years
  OS is defined as the interval from the start of study therapy to death from any cause.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Institute of Hematology and Blood Diseases Hospital at the Chinese Academy of Medical Sciences, Tianjing